CLINICAL TRIAL: NCT00150722
Title: HDL Modulation and Endothelial Function
Brief Title: High-Density Lipoprotein (HDL) Modulation and Endothelial Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Todd Anderson - Principle Investigator, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ethics 18228, TPD 096237; Heart and Stroke Foundation
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2008-11-10 (Estimated); Status verified 2008-11

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis; endothelial function; HDL; Niacin; statins; Stable Atherosclerotic Vascular Disease
MeSH Terms: conditions — Atherosclerosis | interventions — Atorvastatin; Niacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: atorvastatin (or other tolerated statin + Niaspan/placebo) — atorvastatin 80 mg for all, randomized to 1500 mg niacin/placebo and then crossed over

SUMMARY:
It is well known that lowering low-density lipoprotein (LDL) (bad cholesterol) is beneficial for decreasing heart attacks and death. More recently, focus has been on trying to raise HDL (good) cholesterol. The purpose of the present study is to determine if the addition of a sustained release preparation of niacin (Niaspan - a medicine to raise HDL cholesterol) to LDL lowering with a statin type medication results in improved vascular health. The study of the well being of one's vessel wall (endothelial function) will serve as a marker of treatment effect in the study.

Hypotheses: Extended-release (ER) niacin will improve endothelial function measured as brachial flow-mediated dilation (FMD - 10 end-point) and as pulse volume amplitude by pulse arterial tonometry (PAT) (20 end-point) in subjects with established atherosclerosis whose LDL cholesterol is optimally treated with statin therapy.

DETAILED DESCRIPTION:
Purpose: To determine the incremental value of extended-release (ER) niacin in combination with high dose statin therapy on brachial endothelial function in subjects with coronary atherosclerosis.

Hypotheses:

1. ER niacin will improve endothelial function measured as brachial flow-mediated dilation (FMD - primary end-point), hyperemic velocity and as pulse volume amplitude by PAT (20 end-point) in subjects with established atherosclerosis whose LDL cholesterol is optimally treated with statin therapy.
2. Hyperemic pulse volume amplitude in the finger assessed by pulse arterial tonometry (PAT) will correlate with brachial FMD as assessed by high resolution ultrasound of the brachial artery.

Background: In patients with established coronary atherosclerosis, secondary prevention strategies with lipid lowering agents have resulted in event reductions of 25-30%. Despite aggressive cholesterol lowering with statins event rates remain 2-3% per year for subjects at high risk. While many new therapeutic targets have been suggested, recently there has been much interest in modulation of HDL cholesterol. Low HDL is a powerful risk factor for coronary events. HDL functions in the reverse cholesterol transport system to remove excess cholesterol from tissues including the vessel wall. In addition, HDL has other vascular benefits including anti-oxidant and direct endothelial effects. The most effective available way to modulate HDL is with niacin. An ER formulation of niacin (Niaspan - Kos) will be available in Canada in 2005 and has been shown to be efficacious and safe.

The endothelium plays a key role in vascular homeostasis through the release of paracrine factors such as nitric oxide. Dysfunction of the endothelium occurs in response to risk factors and atherosclerosis. Endothelial function can be readily measured non-invasively in humans and pharmacotherapy that has been shown to reduce cardiovascular events improves endothelium-dependent vasodilation. In addition, recent studies have suggested that measures of endothelial function have prognostic implications for subjects at risk for vascular events. As such the measurement of endothelial function has become well established as a surrogate marker of disease activity and will be utilized in the current study. The effect of niacin on endothelial function has not been studied.

Design: The study is a single center, randomized, placebo controlled cross-over design. An open label one month run in phase of atorvastatin therapy will be utilized to establish baseline endothelial function and ensure tolerability of the atorvastatin. Brachial ultrasound determination of FMD and pulse arterial tonometry (PAT) will be utilized. Open label atorvastatin will be continued throughout the study in all subjects. Following baseline measurements of endothelial function, patients will be randomized to placebo or escalating doses of ER niacin for a treatment phase of 3 months. At this point, repeat measurements will be undertaken and subjects will cross-over to the alternate therapy for an additional 3 months followed by final measurements. The use of different methods of endothelial function measurement will allow a comparison of the two.

Subjects will have established coronary atherosclerosis and an HDL < 1.1 mmol/L, and be at least one month post percutaneous coronary intervention (PCI) or 3 months post coronary artery bypass graft (CABG). Exclusion criteria include active gout, gallbladder or peptic ulcer disease, change of endothelial modulating drugs within one month of study initiation or use of niacin.

The primary end-point of the study is brachial artery flow-mediated vasodilation. The primary efficacy analysis will be a comparison of the change in FMD during active ER niacin treatment compared with baseline. The sample size is based on an expected 2% difference in FMD (SD 5%), p <0.05 and power of 80%.

Significance: Despite the reduction of mortality with current LDL lowering approaches, morbidity and mortality remain unacceptably high. HDL has recently gained favor as a therapeutic target to lower cardiovascular event rates. The current study will evaluate the effect of HDL raising on endothelial health, a surrogate marker of atherosclerosis activity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years
* Coronary artery disease

Exclusion Criteria:

* HDL > 1.10 (men), > 1.30 (women)
* PCI within 30 days or CABG within 90 days
* Symptomatic congestive heart failure (CHF)
* Uncontrolled hypertension
* Gout or active gallbladder disease, liver disease or peptic ulcer disease
* Diabetes (or if Fasting blood sugar > 7.0 then hemoglobin A1c [HbA1C] > 6.1 is exclusionary)
* Abnormalities of complete blood count (CBC), creatinine or ALT
* Change in endothelial modulating drugs in the last month or use of niacin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow mediated dilation | 12 weeks

SECONDARY OUTCOMES:
Forearm pulse arterial tonometry (PAT) | 12 weeks
Peak hyperemic velocity | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Todd J Anderson, MD, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Philpott AC, Hubacek J, Sun YC, Hillard D, Anderson TJ. Niacin improves lipid profile but not endothelial function in patients with coronary artery disease on high dose statin therapy. Atherosclerosis. 2013 Feb;226(2):453-8. doi: 10.1016/j.atherosclerosis.2012.10.067. Epub 2012 Nov 5. PMID 23174368